CLINICAL TRIAL: NCT03605628
Title: Influence of Analgesia and Neuromuscular Block on Abdominal Distension and Operating Conditions During Gynecologic Laparoscopic Operations
Brief Title: Influence of Analgesia and Neuromuscular Block on Abdominal Distension and Operating Conditions Laparoscopic Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kreiskrankenhaus Dormagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMB Abdomen
Record Dates: First submitted 2018-04-12; First posted 2018-07-30 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Neuromuscular Blockade

STUDY DESIGN:
Masking Description: Assessment of the quality of operation conditions by the obstretic surgeon without information with regard to the actual depth of the neuromuscular block or the drugs administrated for improvement of the block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- abdominal wall length (Other): Measurement of abdominal wall length during neuromuscular block with a measuring tape
  Interventions: Other: measuring tape; Other: neuromuscular block; Other: Surgical rating score

INTERVENTIONS:
Other: measuring tape — measurement of change in abdominal wall length [cm] during neuromuscular block with a measuring tape.
Other: neuromuscular block — Measurement of the time course of the neuromuscular block: neuromuscular transmission is measured by assessment of the post tetanic count and the train of four ratio using acceleromyography (TOF Watch SX™, Essex Pharma GmbH, Munich, Germany) at the right adductor pollicis muscle with transcutaneous Ag/AgCl electrodes (electrocardiogram electrodes; Ambu Inc., MD 21060 USA);
Other: Surgical rating score — assessment of operating conditions by means of a standardized score: surgical rating score:
  1. extremely poor conditions
  2. poor conditions
  3. acceptable conditions
  4. good conditions
  5. optimal conditions

SUMMARY:
Neuromuscular block improves operation conditions during laparoscopic surgery. In this study, a new measurement tool is assessed: the degree of abdominal distension during the time course of the neuromuscular block is measured and compared with a standardized score (surgical rating score).

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic gynecologic surgery
* American Society of Anesthesiologists Physical Status ASA 1-2

Exclusion Criteria:

* anticipated difficult airway
* increased risk for pulmonary aspiration
* acute infection
* pregnancy
* impaired liver- oder kidney function
* neuromuscular disease
* chronic intake of drugs known to influence neuromuscular blockade

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
change in abdominal wall length (cm) during time course of the block | during operation
  Changes in abdominal wall length are measured during the time course of the neuromuscular block every 15 min.

SECONDARY OUTCOMES:
Change of surgical Rating scale (SRS) scores during neuromuscular block | during operation
  assessment of operating conditions by means of a standardized score: surgical rating score (Martini et al. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs. deep neuromuscular block. Br J Anaesth 2014; 112: 498-505:
  1. extremely poor conditions
  2. poor conditions
  3. acceptable conditions
  4. good conditions
  5. optimal conditions
  The surgical rating score is assessed every 15 min together with abdominal wall length and depth of neuromuscular block
changes of abdominal distension or surgical Rating score (SRS) induced by additional analgesics, sedatives or neuromuscular blocking agents | during operation
  If a bolus of an analgesic, sedative or neuromuscular blocking agent is required because of inadequate anesthesia during the operation, all measurements mentioned above are performed immediately after the injection of the drug in order to assess the effect of the bolus injection.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Soltesz, MD, Principal Investigator — Kreiskrankenhaus Dormagen
Locations (1):
- Kreiskrankenhaus Dormagen, Dormagen, Germany